CLINICAL TRIAL: NCT03992053
Title: The Clinic Application of CBCT XperGuide in Interventional Sacroiliac Joint Pain Therapy
Brief Title: Imaging for SIJ Injection Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects were recruited because of the COVID-19 pandemic. The study is now closed as sponsor milestones (not related to subjects) are completed.
Sponsor: University of Washington (Other)
Collaborators: Philips Medical Systems (Industry)
Responsible Party: Principal Investigator, Jiang Wu, Clinic Assistant Professor, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: STUDY00006861
Record Dates: First submitted 2019-06-07; First posted 2019-06-19 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Sacroiliitis; Sacroiliac Joint Pain
Keywords: 2-dimensional (2-D) fluoroscopy; 3-dimensional (3-D) Computed Tomography (CT) guidance; sacroiliac joint injection
MeSH Terms: conditions — Sacroiliitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): conventional 2-D fluoroscopy guidance as the first choice of guidance
  Interventions: Other: sacroiliac joint injection
- Group 2 (Active Comparator): 3-D CT guidance as the first choice of guidance
  Interventions: Other: sacroiliac joint injection

INTERVENTIONS:
Other: sacroiliac joint injection — Image-guided sacroiliac joint injection under fluoroscopy or CT guidance and the success of intraarticular access was demonstrated by inter-articular contrast spread (the standard of care, not part of study intervention).

SUMMARY:
The Research question: Among two standard image guidance techniques [2-dimension (2-D) conventional Fluoroscopy Versus 3-dimension (3-D) Cone-Beam Computed Tomography (CBCT)], which is the better guidance for Sacroiliac Joint Injection therapy and should be used first?

The specific aims: To detect the difference of the first-time success rate, the cross-over rate, the procedural time, the radiation exposure, the incidence of adverse events/complications, and overall satisfaction score between the 2-D Fluoroscopy versus 3-D CBCT guidance for SIJ injection.

DETAILED DESCRIPTION:
There are no published research studies comparing the injection success rates, procedure duration, radiation exposure, and patient comfort between the two standard imaging systems. The investigators hypothesize that the newer 3-D Cone-beam Based Computer Tomography (CBCT) image system will result in higher success rates, shorter procedure times, fewer image snapshots during the procedure, and less patient discomfort than conventional 2-D fluoroscopy imaging. Although the radiation exposure from one-time low-dose 3-D CT reconstruction with CBCT image system at the beginning of the procedure is higher, the number of later snapshots with the 3-D system is likely to be significantly lower. Therefore the 3-D system may result in overall equivalent radiation exposure to the 2-D system.

A statistical power analysis was conducted and determined that a sample size of 100 (50 per group) will give 80% power for detecting a difference if the true rates are 65% (2-D Fluoroscopy guidance) and 90% (3-D CBCT guidance).

For this study, patients undergoing SIJ injection will be randomized to either Fluoroscopy guidance or CBCT guidance. The primary outcome measure is injection success within 3 attempts of needle placement. Statistical analysis will use the Chi-square test to test whether the rate of injection success differs between the two methods of guidance. In order to provide appropriate clinical care, whenever success is not achieved with the initial guidance method then injection using the other guidance method will be attempted. However, the analysis will only consider whether or not injection success was achieved with the initial guidance method to which the subject was randomized. Whether or not injection success was achieved after crossing over to the other guidance method is not relevant to the primary analysis.

In summary, the investigators would like to formally analyze the differences in these two standard image guidance options in SIJ injection therapy. The investigators propose to randomly select the first imaging system that will be utilized during standard medical care in patients scheduled to undergo an SIJ injection. Presumed that there is a difference in success rate between these two standard images, the imaging procedures are considered to be a part of the research.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and older
2. Clinically diagnosed with sacroiliac joint pain
3. Medically indicated for sacroiliac joint injection (SIJ) therapy (with chronic sacroiliac joint pain, debilitating with pain score > 4 and not responsive to conservative medical management)
4. Financial pre-authorization of SIJ injection approved by insurance
5. English speaking
6. Scheduled for SIJ injection on the Allura machine

Exclusion Criteria:

1. Patient refusal or inability to study informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
The success rate of sacroiliac joint injection | during the procedure periods
  the difference between the success rate of Sacroiliac Joint injection under 3-D CBCT and that of 2-D fluoroscopy guidance
The crossover rate from the first choice guidance to back-up guidance | during the procedure periods
  The crossover rate from the first choice guidance to back-up guidance after three best attempts

SECONDARY OUTCOMES:
Procedure Radiation Dose | during the procedure periods
  Measurement of radiation dose in Rads during procedure.
Procedure Contrast Dose | during the procedure periods
  Measurement of contrast dose in mL during procedure.
Procedure Duration | during the procedure periods
  Length of time for procedure measured in minutes.
Incidence of Treatment-Emergent Adverse Events | during the procedure periods
  Tachycardia, hypertension, vasovagal reaction, procedural abortion, etc.
Procedure Pain | during the procedure periods
  Pre-procedure typical baseline pain and post-procedure typical pain measured on a 0-10 Visual Analog Scale. This scale measures the pain intensity and percentage of pain relief. The left zero end represents no pain and right 10 end represents worst pain imaginable.
Patient Satisfaction Score | during the procedure periods
  Procedure Satisfaction Score measured on a 0-10 Visual Analog Scale. The left zero end represents not satisfied at all and the right 10 end represents 100% satisfaction.
Needle placement attempts | during the procedure periods
  Number of attempts to place needle for procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Wu, MD, Principal Investigator — University of Washington
Locations (1):
- UW Center for Pain Relief, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Patient's IPD is confidential information and well protected under HIPPA law, and reinforced by the Institute IRB policy

REFERENCES:
- [Background] Leschka SC, Babic D, El Shikh S, Wossmann C, Schumacher M, Taschner CA. C-arm cone beam computed tomography needle path overlay for image-guided procedures of the spine and pelvis. Neuroradiology. 2012 Mar;54(3):215-23. doi: 10.1007/s00234-011-0866-y. Epub 2011 Apr 8. PMID 21476020
- [Background] Orth RC, Wallace MJ, Kuo MD; Technology Assessment Committee of the Society of Interventional Radiology. C-arm cone-beam CT: general principles and technical considerations for use in interventional radiology. J Vasc Interv Radiol. 2009 Jul;20(7 Suppl):S538-44. doi: 10.1016/j.jvir.2009.04.026. PMID 19560038
- [Background] Scarfe WC, Farman AG. What is cone-beam CT and how does it work? Dent Clin North Am. 2008 Oct;52(4):707-30, v. doi: 10.1016/j.cden.2008.05.005. PMID 18805225
- [Background] Wagner AL. CT fluoroscopic-guided cervical nerve root blocks. AJNR Am J Neuroradiol. 2005 Jan;26(1):43-4. PMID 15661697
- [Background] Thakor AS, Patel PA, Gu R, Rea V, Amaral J, Connolly BL. MR cone-beam CT fusion image overlay for fluoroscopically guided percutaneous biopsies in pediatric patients. Pediatr Radiol. 2016 Mar;46(3):407-12. doi: 10.1007/s00247-015-3479-5. Epub 2015 Nov 13. PMID 26563298
- [Background] Simopoulos TT, Manchikanti L, Singh V, Gupta S, Hameed H, Diwan S, Cohen SP. A systematic evaluation of prevalence and diagnostic accuracy of sacroiliac joint interventions. Pain Physician. 2012 May-Jun;15(3):E305-44. PMID 22622915
- [Background] Cohen SP, Chen Y, Neufeld NJ. Sacroiliac joint pain: a comprehensive review of epidemiology, diagnosis and treatment. Expert Rev Neurother. 2013 Jan;13(1):99-116. doi: 10.1586/ern.12.148. PMID 23253394
- [Background] King W, Ahmed SU, Baisden J, Patel N, Kennedy DJ, Duszynski B, MacVicar J. Diagnosis and treatment of posterior sacroiliac complex pain: a systematic review with comprehensive analysis of the published data. Pain Med. 2015 Feb;16(2):257-65. doi: 10.1111/pme.12630. PMID 25677327
- [Background] Kennedy DJ, Engel A, Kreiner DS, Nampiaparampil D, Duszynski B, MacVicar J. Fluoroscopically Guided Diagnostic and Therapeutic Intra-Articular Sacroiliac Joint Injections: A Systematic Review. Pain Med. 2015 Aug;16(8):1500-18. doi: 10.1111/pme.12833. Epub 2015 Jul 14. PMID 26178855
- [Background] Kasliwal PJ, Kasliwal S. Fluoroscopy-Guided Sacroiliac Joint Injection: Description of a Modified Technique. Pain Physician. 2016 Feb;19(2):E329-38. PMID 26815260
- [Background] Hawkins CM, Kukreja K, Singewald T, Minevich E, Johnson ND, Reddy P, Racadio JM. Use of cone-beam CT and live 3-D needle guidance to facilitate percutaneous nephrostomy and nephrolithotripsy access in children and adolescents. Pediatr Radiol. 2016 Apr;46(4):570-4. doi: 10.1007/s00247-015-3499-1. Epub 2015 Dec 4. PMID 26637320